CLINICAL TRIAL: NCT05651074
Title: A Pharmacokinetic/Pharmacodynamic Study to Evaluate the Effect of Omeprazole of Vicagrel in Healthy Subjects
Brief Title: Assessment of the Effect of Omeprazole on Vicagrel in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCP1-Ⅰ-07
Record Dates: First submitted 2022-11-17; First posted 2022-12-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — methyl 2-(2-acetoxy-6,7-dihydrothieno(3,2-c)pyridin-5(4H)-yl)-2-(2-chlorophenyl)acetate; Omeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vicagrel and omeprazole (Experimental): D1 single dose of vicagrel was administered. Omeprazole administration was started on D4, once daily for 5 days, and a single dose of vicagrel and omeprazole coadministration on day 9.
  Interventions: Drug: Vicagrel and omeprazole

INTERVENTIONS:
Drug: Vicagrel and omeprazole — 18 mg vicagrel capsules and 40 mg omeprazole magnesium enteric-coated tablets

SUMMARY:
The primary objective of the study is to evaluate the effects of omeprazole on the PK and PD of a single dose of vicagrel in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent before study, and fully understand the study content, process and possible adverse reactions;
2. Able to complete the study in compliance with the protocol;
3. Subject (including partner) is willing to voluntarily take effective contraceptive measures from screening through 6 months after the last dose of study drug (see Appendix 5 for details);
4. Male and female subjects between the ages of 18 and 45 years, inclusive;
5. At least 50 kg for male subjects, 45 kg for female subjects, with a Body Mass Index (BMI= Weight/Height2) between 18-28 kg/m2, inclusive;
6. With normal or clinically insignificant abnormal results of physical examination and vital signs test;
7. CYP2C19 normal metabolizers (CYP2C19*1/*1).

Exclusion Criteria:

1. More than 5 cigarettes per day on average within 3 months before the study;
2. History of sensitivity to drugs similar to the study drug or have high sensitivity to clopidogrel, or hypersensitivity to omeprazole, other benzimidazoles, or any excipients, allergic constitution (e.g. allergy to various drugs and foods);
3. History of drug abuse, drug use, alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL beer, 25 mL spirit or 100 mL wines);
4. Donation or loss of a significant volume of blood (> 450 mL) within 3 months prior to screening;
5. Intake of any prescription drugs, over-the-counter drugs, vitamin or herbal medicine within 14 days prior to receiving study drug;
6. Consumption of any special diet (such as grapefruit, pitaya, mango, pomelo, etc.) or subjects have engaged strenuous exercise or any other factors affecting drug absorption, distribution, metabolism and excretion within 14 days prior to receiving study drug;
7. Intake of any drug which Have taken strong inhibitors and/or inducers of liver metabolic enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4 and 3A5) within 28 days before the first medication, and strong inhibitors of liver metabolic enzymes such as: ciprofloxacin, clopidogrel, Itraconazole, ketoconazole, ritonavir, troleandomycin, etc., strong inducers of liver metabolism enzymes such as: rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc. (For details see Appendix 6);
8. Recent major changes in diet or exercise habits;
9. Use of an investigational drug or product, or participation in a drug research study within 3 months prior to receiving study drug;
10. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption;
11. Suffering from any diseases that may increase the risk of bleeding, such as hemorrhoids, acute gastritis, stomach and duodenal ulcers, Thrombocytopenic Purpura and hemophilia, etc;
12. Family history of coagulation or bleeding disorders (e.g., hemophilia)/symptoms (e.g., vomiting blood, black stools, severe or recurrent nosebleeds, coughing up blood, significant hematuria, or intracranial hemorrhage) or suspected vascular malformations, such as aneurysms or early onset strokes, in the individual or in their immediate family;
13. A clinically significant 12-lead ECG abnormality;
14. Positive test results of blood pregnancy or subject is lactating for female subjects;
15. Any clinically significant abnormalities/findings in laboratory tests, or any clinically significant disease including but not limited to gastrointestinal, renal, hepatic, neurological system, blood, endocrine, tumor, lung, immune, mental, or cardiovascular and cerebrovascular diseases;
16. Positive test results for viral hepatitis (including hepatitis B and C), HIV antibody or syphilis antibody;
17. Acute illness or concomitant medication from screening to the first dosing of study medication;
18. Consumption of chocolate or any food or beverages containing caffeine or (rich containing) xanthine within 48 h prior to receiving the first dosing of study medication;
19. Consumption of any product containing alcohol within 24 h prior to receiving the first dosing of study medication, or positive results from a screen for alcohol;
20. Positive results from a screen for urine drug test (Morphine, marijuana);
21. Subjects were vaccinated within 4 weeks prior to screening, or planned to be vaccinated during the trial;
22. Any condition which in the opinion of Investigator is not suitable for subjects to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation [IPA] evaluated in healthy subjects to treatment with vicagrel | Day 2 of each period
Platelet reactivity index [PRI] evaluated in healthy subjects to treatment with vicagrel | Day 2 of each period
maximum plasma concentration (Cmax) | Up to 48 hours postdose on Day 3 for each period
Area under the concentration-time curve (AUC) | Up to 48 hours postdose on Day 3 for each period

SECONDARY OUTCOMES:
Assess the safety of a single dose of vicagrel and a combination of vicagrel and omeprazole in healthy subjects by assessment of adverse events and symptoms and physical examination, clinical laboratory tests, vital signs,12-ECG. | Day1-Day11

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Center of The First Hospital of Jilin University, Changchun, Jilin, China